CLINICAL TRIAL: NCT00122512
Title: Phase 2a Study of Tenofovir Disoproxil Fumarate (TDF) for Prevention of HIV - An Extended Safety Evaluation
Brief Title: Study of Tenofovir Disoproxil Fumarate (TDF) for Prevention of HIV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: FHI 360 (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 9876
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2006-02-10 (Estimated); Status verified 2006-02

CONDITIONS: HIV Infections
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU international units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; TDF tenofovir disoproxil fumarate, GS-4331-05, PMPA prodrug; µg microgram; ULN upper limit of the normal range; WB Western Blot; Human Immunodeficiency Virus; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate

SUMMARY:
This Phase 2a study involving Tenofovir Disoproxil Fumarate (TDF) will provide extended safety data for high-risk men. Secondarily, the study will assess the feasibility of conducting the trial and evaluate the preliminary effectiveness of TDF 300 mg as an HIV prevention method when taken once a day.

DETAILED DESCRIPTION:
TDF has been selected for investigation as prophylaxis against HIV in high-risk men because of its unique pharmacologic profile. In addition to the convenience of being a once daily single tablet, TDF's safety profile is comparable to placebo among HIV infected persons, it has striking anti-HIV potency, and it has low potential for selection of resistant viruses. TDF is cleared from the body by the kidneys and is not metabolized by the liver. Therefore, TDF has limited potential to have pharmacokinetic interactions with other hepatically metabolized drugs. Each of these properties is necessary given the realities of the intended target populations. Moreover, initial prevention studies in simian models have provided encouraging results. Finally, the drug's sponsor is supportive of investigating the potential use of TDF as a preventive, as well as therapeutic agent, will provide TDF for the study, and is willing to make a good faith effort to make TDF available for public health use should it prove to be effective for HIV prevention.

ELIGIBILITY:
* Be willing and able to give informed consent
* Be 18 years or older
* Be willing to use study product as directed
* Be willing to adhere to follow-up schedule
* Be willing to participate in the study for up to 12 months
* Be in general good health (no active, serious infections that require parenteral antibiotics, no active clinically significant medical conditions, including heart disease, diabetes, asthma, alcoholism, and cancer)
* Meet at least one of these three high risk criteria: *Sex with sex worker/bar girl in last 3 months;

  * Sex with 2 or more women in last 3 months;
  * Sexually transmitted disease (STD) in last 3 months
* Have absence of HIV antibodies by rapid test (at screening and enrollment visit)
* Have absence of hepatitis B (HB) surface antigen (sAg)
* Have adequate renal function (serum creatinine <1.5 mg/dL)
* Have adequate liver function (hepatic transaminases (ALT <54 U/L and AST<46 U/L)
* Have adequate serum phosphorus (>2.2 mg/dL)
* Not be intending to relocate out of the area for the duration of the study participation and does not have a job or other obligations that may require long absences from the area
* Not be receiving an experimental HIV vaccine

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500

PRIMARY OUTCOMES:
To evaluate the extended safety of TDM 300mg daily among HIV-uninfected men

SECONDARY OUTCOMES:
To evaluate the feasibility (i.e. accrual, retention, adherence, change in behavior) of conducting a large scale trial of TDF for HIV prevention in men recruited from a resource-limited setting
To assess the preliminary effectiveness of TDF in preventing HIV infection among men at high risk for HIV

CONTACTS AND LOCATIONS:
Overall Officials: Irving Hoffman, PA, MPH, Principal Investigator — UNC Center for Infectious Diseases
Locations (1):
- UNC Project, Kamuzu Central Hospital, Lilongwe, Malawi